CLINICAL TRIAL: NCT03156374
Title: Proof of Concept Study To Assess Women's Likability and Stress in Timing Frozen Embryo Transfer by Following Two Different Methods
Brief Title: Timing Frozen Embryo Transfer by Following Two Different Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROTOCOL-0897
Record Dates: First submitted 2017-04-28; First posted 2017-05-17 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Intervention Model Description: Parallel use of ovulation test and standard hospital monitoring, for agreement of methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovulation test use (Experimental): Use of both ovulation tests and standardised care
  Interventions: Device: Test use

INTERVENTIONS:
Device: Test use — Use of home ovulation test to predict ovulation

SUMMARY:
This proof of concept study is designed to determine the practicality of using home ovulation tests to enable optimum timing for transfer of frozen embryos in a natural menstrual cycle in comparison to the standard ultrasound and serum monitoring currently conducted by many IVF clinics.

DETAILED DESCRIPTION:
The study will evaluate the ability of home ovulation tests to accurately time Frozen Embryo Transfer (FET) directly compared to standard clinical procedures. In addition, women's likability and stress associated with timing a FET cycle using both methods will be evaluated by collecting qualitative data using standardised questionnaires.

The impact of psychological stress on FET outcome such as implantation rates and viability at first scan will be considered in order to gather information for the design of a larger clinical study and basic financial data will also be collected, in order to pilot a cost-effectiveness evaluation of the two FET timing methods.

A subset of volunteers will collect daily urine samples from day after embryo transfer until confirmation of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 24 to 45 years of age
* Undergoing no more than 5frozen embryo transfer
* Average cycle length between 26 and 35 days
* Willing to provide written informed consent to participate in the study and comply with all study procedures

Exclusion Criteria:

* More than five IVF frozen embryo cycle
* Undergoing FET following cancer treatment
* Self-reported drug or alcohol dependency
* Self-reported history of depression, anxiety and panic attacks

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological women only
Enrollment: 46 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers where ADOT use enables equivalent timing of FET compared to clinic visit | 9 months
  Examination as to whether using ADOT would have enabled correct timing of FET when compared to clinic visit

SECONDARY OUTCOMES:
Measurement of women's psychological distress | 9 months
  Use of validated questionnaire to assess stress level
Positive and negative experience in using ovulation tests in FET | 9 months
  Qualitative assessment of women's FET treatment experience when using ADOT compared to standard clinical procedures during the study via a semi-structured interview following embryo transfer
FET success | 9 months
  Implantation rate

CONTACTS AND LOCATIONS:
Locations (1):
- IVFAustralia - Bondi Junction, Bondi Junction, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No